CLINICAL TRIAL: NCT06749119
Title: Effect of Age on Recipient Site Wound Healing in Free Gingival Graft Operation
Brief Title: The Effects of Age on Wound Healing on Free Gingival Graft Surgery in the Treatment of Attached Keratinized Gingival Deficiency by Determining Clinical and Biochemical Outcomes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 09.2020.660
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-11

CONDITIONS: Wound Healing; Tissue Grafts; Age; Vegf; TGF-β

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Young group: Aged 20-35 years (Active Comparator): They received free gingival operation. Graft was harvested from palatal region and placed to the recipient site. Wound fluid samples were collected from 4 regions of the wound at baseline, 4-,7-,14-days. Clinical measurements were done at baseline, 1-,3-,6-months postoperatively.
  Interventions: Procedure: Free gingival graft operation
- Adult group: Aged 50-65 years (Active Comparator): They received free gingival operation. Graft was harvested from palatal region and placed to the recipient site. Wound fluid samples were collected from 4 regions of the wound at baseline, 4-,7-,14-days. Clinical measurements were done at baseline, 1-,3-,6-months postoperatively.
  Interventions: Procedure: Free gingival graft operation

INTERVENTIONS:
Procedure: Free gingival graft operation — Free gingival graft was harvested from palatal region and stabilized on the maxillary anterior recipient bed with sutures .

SUMMARY:
This study aimed to assess the effects of age on wound healing on free gingival graft (FGG) surgery in the treatment of attached keratinized gingival deficiency by determining clinical and biochemical outcomes.

DETAILED DESCRIPTION:
Aim of this study was to evaluate the effect of age on clinical and biochemical healing outcomes on FGG surgery in the treatment of attached keratinized gingival deficiency (≤2 mm) at mandibular anterior region. A total of 30 systemically healthy patients, divided into two groups and planned for FGG operations, were included in this study. These groups are; Group l : 15 patients in the age range of 20-35, group 2: 15 patients in the age range of 50-65. Gingival crevicular fluid and wound fluid samples were taken from these patients to analyze VEGF, EGF and TGF-B1 levels by ELISA. Wound fluid samples were taken baseline, 4,7, and 14 days after surgery.

Clinical parameters included measurement of probing depth (PD), clinical attachment level (CAL), bleeding of probing (BOP), plaque index (PI), gingival index (GI) at 6 sites per tooth except the third molars were measured at baseline and l, 3 and 6 months after surgery. Keratinized gingiva width, keratinized gingiva thickness of the operation sites were measured baseline and 1,3 and 6 months after surgery. Vertical dimension of the graft, horizontal dimension of the graft, graft thickness were measured at baseline and 1,3,6 months after surgery. Graft area measurements were calculated on standard photographs by a Java-based analysis program (ImageJ, National Institutes of Health, Bethesda, MD) to determine the shrinkage rate of the grafts. The graft shrinkage ratio was calculated as the difference between baseline to 1-month, baseline to 3-months, baseline to 6-month graft site value. Data were analyzed using appropriate statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* having ≤2mm of keratinized gingiva in at least 1 mandibular anterior tooth
* periodontally healthy with full-mouth bleeding and plaque score ≤ 10%
* no use of any drugs that will affect periodontal tissue health and healing process
* absence of any systemic condition or illness

Exclusion Criteria:

* smokers
* previous periodontal surgery
* a pathology in the apical region of the tooth
* pregnancy, lactation

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-04-14 (Actual); Primary Completion 2024-12-27 (Estimated); Study Completion 2024-12-27 (Estimated)

PRIMARY OUTCOMES:
Shrinkage percentage (%) | from baseline to 1-,3-,6- months
  Shrinkage percentage of the graft area due to the changes in graft dimensions

SECONDARY OUTCOMES:
VEGF levels (pg/ml) | from baseline to 1-,3-,6- months
  change in wound fluid VEGF levels from baseline to 1-,3-,6- months after surgery
EGF levels (pg/ml) | baseline to 1-,3-,6- months
  change in wound fluid EGF levels from baseline to 1-,3-,6- months after surgery
TGFβ-1 levels (pg/ml) | from baseline to 1-,3-,6- months
  change in wound fluid TGFβ-1 levels from baseline to 1-,3-,6- months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No